CLINICAL TRIAL: NCT06218862
Title: Clinical Effects of Sivelestat Sodium on Improving ARDS in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: liyuting@jlu.edu.cn
Record Dates: First submitted 2024-01-22; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: ARDS Due to Disease Caused by SARS Co-V-2
MeSH Terms: interventions — Antiviral Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sivelestat sodium: Sivelestat sodium was administered through a 24-hour continuous intravenous infusion at a rate of 0.2 mg/kg/h, for a maximum duration of 14 days.
  Interventions: Drug: Sivelestat sodium
- Control: Not use Sivelestat sodium
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Sivelestat sodium — Sivelestat sodium was administered through a 24-hour continuous intravenous infusion at a rate of 0.2 mg/kg/h, for at least 72 hours and a maximum duration of 14 days.
  Other Names: antiviral
  Groups: Sivelestat sodium
Drug: Control — Not use Sivelestat sodium
  Other Names: antiviral
  Groups: Control

SUMMARY:
The goal of this retrospective multicentre cohort study is to examine the association between receipt of sivelestat and improvement in oxygenation among patients with acute respiratory distress syndrome (ARDS) induced by COVID-19. We used propensity score matching to compare the outcomes of patients treated with sivelestat to those who were not. The primary outcome was the PaO2/FiO2 ratio on Day 3. Secondary outcomes included 28-day mortality, alive and ICU-free days within 28 days, non-mechanical ventilation time within 28 days, the lengths of stay in the ICU and hospital, proportion of patients requiring extracorporeal membrane oxygenation (ECMO), proportion of patients undergoing endotracheal intubation or tracheotomy, and incidence of adverse events (AEs) or severe adverse events (SAEs).

DETAILED DESCRIPTION:
We conducted a retrospective cohort study of patients admitted between December 2022 and May 2023 to general ICUs, respiratory ICUs and emergency ICUs across 14 hospitals in Jilin Province, China. We used propensity score matching to compare the outcomes of patients treated with sivelestat to those who were not. Sivelestat sodium was administered through a 24-hour continuous intravenous infusion at a rate of 0.2 mg/kg/h, for a maximum duration of 14 days.The primary outcome was the PaO2/FiO2 ratio on Day 3. Secondary outcomes included 28-day mortality, alive and ICU-free days within 28 days, non-mechanical ventilation time within 28 days, the lengths of stay in the ICU and hospital, proportion of patients requiring extracorporeal membrane oxygenation (ECMO), proportion of patients undergoing endotracheal intubation or tracheotomy, and incidence of adverse events (AEs) or severe adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

1) equal to or more than 18 years old, 2) had positive COVID-19 reverse transcriptase-polymerase chain reaction test results from upper airway swab, 3) fulfilled the Berlin definition of ARDS

Exclusion Criteria:

pregnant or lactating women, those with concomitant severe chronic respiratory diseases or end-stage malignant tumours, patients with duration of hospital stay or sivelestat administration less than 72 hours and patients for whom complete outcome data were not available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We conducted a retrospective cohort study of patients admitted between December 2022 and May 2023 to general ICUs, respiratory ICUs and emergency ICUs across 14 hospitals in Jilin Province, China.
Sampling Method: Probability Sample
Enrollment: 387 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio on Day 3. | 3 days
  PaO2/FiO2 ratio on Day 3.

SECONDARY OUTCOMES:
28-day mortality | 28 days
  28-day mortality
non-mechanical ventilation time within 28 days | 28 days
  non-mechanical ventilation time within 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Yuting Li, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- Yuting Li, Changchun, None Selected, China